CLINICAL TRIAL: NCT00068952
Title: A Phase III, Randomized, Open-Label Study Of IV Edotecarin Vs Temozolomide Or Carmustine (BCNU) Or Lomustine (CCNU) In Patients With Glioblastoma Multiforme At First Relapse After Alkylator-Based (NEO) Adjuvant Chemotherapy
Brief Title: Study of IV Edotecarin Vs Temozolomide or Carmustine (BCNU) or Lomustine (CCNU) in Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDOAGL-8725-001; A5921009
Record Dates: First submitted 2003-09-12; First posted 2003-09-16 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — edotecarin; Temozolomide; Carmustine; Lomustine

INTERVENTIONS:
Drug: Edotecarin
Drug: Temozolomide
Drug: Carmustine (BCNU)
Drug: Lomustine (CCNU)

SUMMARY:
The purpose of this clinical trial is to study Edotecarin in patients with the brain tumor glioblastoma multiforme (GBM) who have progression or first recurrence following initial treatment with surgery, radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have biopsy-proven GBM. First relapse (progression or recurrence) of GBM after surgery (or biopsy) and treatment with radiotherapy (conventional fractionated external beam) and chemotherapy (temozolomide- or nitrosurea-based therapy)
* Must have past biopsy samples available for central pathology review
* Must have evidence on Gd-MRI of progressive/recurrent disease
* Must have measurable disease on Gd-MRI obtained within 14 days prior to start of study treatment
* Must be at least 18 years of age
* Must have a Karnofsky Performance Status score of at least 70
* If being treated with steroids, the steroid dose must be stable or decreasing for 1 week prior to randomization
* If being treated with anticonvulsants, must have no change in the type of anticonvulsants for 2 weeks prior to randomization
* All acute toxic effects (except for alopecia) of any prior treatment must have resolved or are no greater than grade 1 (NCI Common Toxicity Criteria, Version 2.0)
* Baseline laboratory data must be within the following limits: absolute neutrophil count at least 1500; platelets at least 100,000; hemoglobin at least 9.0 g/dL; serum creatinine no greater than 1.5 mg/dL, total serum bilirubin no greater than 1.5 times the upper limit of the normal range; SGOT and SGPT no greater than 2.5 times the upper limit of the normal range; albumin at least 3.0 g/dL, serum or urine pregnancy test (for females of childbearing potential) negative within 7 days prior to start of study treatment
* At least 6 weeks must have elapsed since completion of prior nitrosurea therapy; at least 4 weeks since completion of prior temozolomide therapy
* Must have written informed consent
* Must be able and willing to comply with study procedures
* 	Must have received prior treatment with radiotherapy (conventional fractionated external beam) and (neo)adjuvant/concurrent chemotherapy (with a temozolomide- or a nitrosurea-based containing )regimen for GBM

Exclusion Criteria:

* Must not have received prior treatment (except for surgical debulking) of first relapse (progression or recurrence) of GBM
* Must not have received prior treatment with another topoisomerase-I inhibitor (e.g. irinotecan, topotecan, rubitecan)
* Must not have had radiosurgery or radiotherapy within 1 month prior to randomization
* Must not have had prior brachytherapy or chemotherapy wafer implantation
* Must not have had prior high-dose chemotherapy with bone marrow or stem cell support
* Must not receive concomitant treatment with any other investigational agent or anti-cancer treatment during the study
* Must not be currently enrolled in another therapeutic clinical trial for the treatment of GBM
* Must not currently (or in the past 5 years) have other malignancies (except for adequately treated basal cell or squamous cell skin cancer or non-invasive cervical cancer)
* Must not have any of the following in the past 6 months: myocardial infarction (heart attack), severe/unstable angina, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident (stroke), or transient ischemic attack (TIA)
* Must not have had any of the following in the past 2 months: pulmonary embolus (blood clot in lungs), deep venous thrombosis (blood clot in veins), or other significant thromboembolic event
* Must not have an ongoing cardiac dysrhythmia (abnormal heart rhythm) of grade 2 or higher (NCI Common Toxicity Criteria, Version 2.0)
* Must not have known human immunodeficiency virus (HIV) infection
* Must not be pregnant or breastfeeding. Patients (male and female) must be surgically sterile (or postmenopausal for females) or must agree to use effective contraception during the period of study treatment
* Must not be inappropriate for entry into the study, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Start 2003-08; Study Completion 2006-03

PRIMARY OUTCOMES:
To compare the overall survival associated with edotecarin versus that associated with temozolomide or BCNU or CCNU for the treatment of patients with GBM at first relapse previously treated with alkylator-based (neo)adjuvant therapy

SECONDARY OUTCOMES:
To assess measures of tumor control To evaluate measures of clinical benefit To assess the safety profile of edotecarin To assess the PK profile of edotecarin and the potential for drug interactions between anticonvulsants and edotecarin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (19):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evanston, Illinois
  - Pfizer Investigational Site, Edgewood, Kentucky
  - Pfizer Investigational Site, Edgweood, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, Summit, New Jersey
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
- Australia (3):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, East Bentleigh, Victoria
  - Pfizer Investigational Site, Clayton
- Austria (2):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Vienna
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Croatia (2):
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Zagreb
- Czechia (2):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- France (2):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Nantes Saint Herblain
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Regensburg
  - Pfizer Investigational Site, Tübingen
- Pfizer Investigational Site, Bangalore, India
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Padua
- Pfizer Investigational Site, Moscow, Russia
- South Africa (2):
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Pretoria
- Spain (3):
  - Pfizer Investigational Site, Badalona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat
  - Pfizer Investigational Site, Oviedo
- Pfizer Investigational Site